CLINICAL TRIAL: NCT03317574
Title: A Randomized, Double-blind, Active Drug Controlled, Multi-center, Phase Ⅰ/Ⅲ Study to Determine the Efficacy and Safety of Meditoxin® in Treatment of Crow's Feet Line
Brief Title: MEDITOXIN® in Treatment of Crow's Feet Line
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT01-KR17CFL903
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Crow's Feet Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MEDITOXIN (Experimental)
  Interventions: Drug: botulinum toxin type A
- BOTOX (Active Comparator)
  Interventions: Drug: botulinum toxin type A

INTERVENTIONS:
Drug: botulinum toxin type A — 24 units botulinum toxin Type A (total dose) injected into bilateral Crow's Feet Line areas
  Other Names: MEDITOXIN
  Arms: MEDITOXIN
Drug: botulinum toxin type A — 24 units botulinum toxin Type A (total dose) injected into bilateral Crow's Feet Line areas
  Other Names: BOTOX
  Arms: BOTOX

SUMMARY:
to determine the efficacy and safety of Meditoxin® in treatment of crow's feet line

ELIGIBILITY:
Inclusion Criteria:

* Male or female of at least 20 to 65 years old
* Bilaterally symmetrical moderate-to-severe CFL at maximum smile on the FWS as rated by the investigator

Exclusion Criteria:

* Diagnosis of myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis
* Patients with allergy or hypersensitivity to the investigational drugs or their components
* Patients who have bleeding tendency or taking anti-coagulant
* Female subjects who are pregnant or lactating. Female subjects of childbearing age who have a plan to get pregnant during the study period, or do not use available contraceptive methods (Women of childbearing age should have negative urine pregnancy test results at baseline visit (0 week) prior to the first injection.)
* Patients who are participating in other clinical trials or have participated in other clinical trials 30 days before screening
* Patients who are unable to communicate or follow the instructions
* Patients who are not eligible for this study based on the judgment of an investigator

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-05-14 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving None or Mild on the Investigator's Assessment of the Severity of Crow's Feet Lines (CFL) at Maximum Smile Using the Facial Wrinkle Scale(FWS) | 4 weeks
  The Investigator assessed the severity of the patient's Crow's Feet lines at maximum smile using the 4-point Facial Wrinkle Scale where 0=none, 1=mild, 2=moderate or 3=severe. The percentage of participants with a score of none or mild at Day 30 is reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Gyeonggi-do, South Korea